CLINICAL TRIAL: NCT04319484
Title: A Randomized Controlled Study of Lenvatinib Following Liver Transplantation in Patients of Hepatocellular Carcinoma With Portal Vein Tumor Thrombus
Brief Title: Lenvatinib Following Liver Transplantation in Patients of Hepatocellular Carcinoma With Portal Vein Tumor Thrombus
Acronym: LLTHVV
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Renji8791
Record Dates: First submitted 2020-01-19; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Hepatocellular Carcinoma; Portal Vein Tumor Thrombus; Liver Transplantation
Keywords: Liver Transplantation; Hepatocellular Carcinoma; Portal Vein Tumor Thrombus; Lenvatinib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Intervention Model Description: Patients enrolled in the study were randomly allocated in the lenvatinib group (54 patients) and the control group (54 patients) after stable condition.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- lenvatinib (Experimental): Patients in the lenvatinib group are given lenvatinib within 1-2 months after operation (dose: body weight < 60 kg: 8 mg/day, body weight ≥ 60 kg 12 mg/day).
  Interventions: Drug: lenvatinib
- Placebo (Placebo Comparator): The placebo pills are made identical to the investigating lenvatinib in appearance
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lenvatinib — 1-2 months after liver transplantation, participants are given lenvatinib with an initial dose of 8 mg (body weight < 60 kg) or 12 mg orally once a day. The initial dose was 8 mg (body weight < 60 kg) or 12 mg orally once a day.
  Other Names: experiment
  Arms: lenvatinib
Drug: Placebo — 1-2 months after liver transplantation, participants are given Placebo with an initial dose of 8 mg (body weight < 60 kg) or 12 mg orally once a day. The initial dose was 8 mg (body weight < 60 kg) or 12 mg orally once a day.
  Other Names: Control
  Arms: Placebo

SUMMARY:
The aim of this study is to observe the efficacy and safety of lenvatinib in preventing recurrence of hepatocellular carcinoma patients with portal vein tumor thrombus after liver transplantation.

DETAILED DESCRIPTION:
The research is an open, randomized, single-center study. Patients of hepatocellular carcinoma with portal vein cancer thrombus who underwent liver transplantation are included according to the criteria of admission. After operation, the regimen of calcineurin inhibitors, mycophenolate mofetil, sirolimus or everolimus with glucocorticoids removed at an early stage are used. Patients enrolled in the study were randomly allocated in the lenvatinib group (54 patients) and the control group (54 patients) after stable condition. Patients in the control group are given supportive treatment and regular follow-up. Patients in the lenvatinib group are given lenvatinib within 1-2 months after operation (dose: body weight < 60 kg: 8 mg/day, body weight ≥ 60 kg 12 mg/day). The baseline data of patients are collected before allocation. Serum and imaging examination are checked regularly every month to monitor the recurrence of hepatocellular carcinoma and the side effects of lenvatinib. The efficacy and safety of lenvatinib in patients of hepatocellular carcinoma with portal vein tumor thrombus are observed, and the clinicopathological factors affecting the efficacy of lenvatinib are analyzed. When side effects of lenvatinib occur, the dosage can be reduced according to the patients' condition until discontinuation. When tumor recurrence occurs, a multidisciplinary team will draw up specific treatment plans according to the patients' condition, including surgical resection, interventional therapy, radiofrequency therapy, radiotherapy and targeted therapy (Patients in the control group can add lenvatinib, and patients in the lenvatinib group can decide whether to continue using it according to the patients' condition).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent liver transplantation were preoperatively imaging diagnosed as hepatocellular carcinoma with portal vein tumor thrombus.
2. Male or female patients aged 18 to 75.
3. ECOG physical condition was 0-2 points.
4. Child-Pugh A grade of liver function.
5. Targeted therapy is acceptable within 1-2 months after liver transplantation.
6. Immunosuppressive regimen consists of calcineurin inhibitor, mycophenolate mofetil and sirolimus.
7. No history of surgical resection of liver tumors and targeted drug therapy before liver transplantation.
8. Good liver, kidney and bone marrow function: serum albumin > 28g/L, total bilirubin ≤ 3 mg/dL (51.3 umol/l), ALT and AST ≤ 5 times the upper limit of normal range; serum creatinine ≤ 1.5 times the upper limit of normal range; hemoglobin > 90 g/L, neutrophil count (ANC) > 1.5 * 10 ^ 9/L, platelet count > 60 * 10 ^ 9/L; PT-INR < 2.3, or PT within 6 seconds over normal upper limit.
9. For fertile female patients, the serum/urine pregnancy test should be negative within 7 days before treatment.
10. All male and female participants must take reliable contraceptive measures during the trial and within four weeks after the end of the trial.
11. The participants have the capability of oral medication.
12. The participants must sign the consent form.

Exclusion Criteria:

1. Hepatocellular carcinoma with invasion of hepatic vein and inferior vena cava
2. Life expectancy is less than 3 months
3. The recurrence and metastasis of hepatocellular carcinoma are highly suspected.
4. Patients are with other malignant tumors simultaneously.
5. Patients are anaphylaxis to the inactive ingredients of lenvatinib or drugs.
6. Pregnant or lactating women (Female participants need pregnancy test within 7 days before treatment).
7. Preoperative history of severe cardiovascular disease: congestive heart failure > NYHA grade 2; active coronary heart disease (myocardial infarction occurred within 6 months before entry into the study); severe arrhythmia requiring antiarrhythmic treatment (allowable use of beta-blockers or digoxin); uncontrolled hypertension.
8. History of HIV infection.
9. Severe clinical active infections (> NCI-CTCAE version 3.0).
10. Epilepsy patients requires medication (e.g. steroids or antiepileptic drugs).
11. Patients with kidney diseases requires renal dialysis.
12. Drug abuse, medical symptoms, mental illness or social status that may interfere with participants'participation in research or evaluation of research results.
13. Patients who could not swallow oral drugs, such as those with severe upper gastrointestinal obstruction and need gastric tube feeding.
14. Other anti-angiogenesis therapies, surgery, TACE, local therapy and systemic chemotherapy were given before the treatment after liver transplantation.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2020-05-02 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
3 years recurrence-free survival rate | 3 years
  Tumor-free survival in 3 years

SECONDARY OUTCOMES:
1 year recurrence-free survival rate | 1 years
  Tumor-free survival in 1 years
1 year overall survival rate | 1 year
  Overall survival refers to the time from treatment to death for any reason.
3 years overall survival rate | 3 years
  Overall survival refers to the time from treatment to death for any reason.
5 years overall survival rate | 5 years
  Overall survival refers to the time from treatment to death for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: qiang xia, doctor, Study Chair — RenJi Hospital

IPD SHARING:
Plan to Share IPD: No